CLINICAL TRIAL: NCT00648284
Title: An Observational Study to Assess the Impact of Pharmacological Intervention and Life Style Changes in the Reduction of Cardiovascular Disease in Patients With Diabetes Type 2 in Greece
Brief Title: Cardiovascular (CV) Risk Evaluation In Type 2 Diabetes Subjects
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Other Study IDs: 104243; Avandia OB
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Type 2 Diabetes Mellitus; CV Risk
Keywords: Type 2 diabetes; CV risk; rosiglitazone; AVANDIA
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The primary objective of this study is to assess the total CV risk in patients with type 2 diabetes and also to assess the impact of rosiglitazone in the total CV risk and the parameters of metabolic syndrome.

ELIGIBILITY:
Inclusion criteria:

* Patients with diabetes type 2 that their physician has decided to prescribe AVANDIA for better control of their condition
* Have signed informed consent

Exclusion Criteria:

* Patients with ALT > 2.5x the normal value
* With heart failure symptoms
* With diagnosis of angina pectoris or stable angina demanding continuous treatment with nitrates
* With recent myocardial infarction (<6 months)
* With severe renal disfunction
* Pregnant or lactating or planned to be pregnant during the study
* Under investigational drug treatment
* Alcoholic or drug abuser

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100
Dates: Start 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline